CLINICAL TRIAL: NCT07289334
Title: Tenotomy Versus no Tenotomy of the Long Head of the Biceps in Rotator Cuff Repair: Clinical-functional Analysis and Ultrasound Evaluation
Brief Title: Tenotomy Versus no Tenotomy LHB in Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Josep Maria Mora Guix, Surgeon of Shoulder Unit, Consorci Sanitari de Terrassa, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-14-105-018
Record Dates: First submitted 2025-09-30; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Long Head of Biceps Brachii Lesions; Rotator Cuff Tears
Keywords: long head biceps; rotator cuff tears; tenotomy; no tenotomy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to two groups, TENOTOMY (n=25) and NO TENOTOMY (n=29), using a centralized random number program.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NO TENOTOMY (Placebo Comparator): NO TENOTOMY OF LHBT + ROTATOR CUFF REPAIR
  Interventions: Procedure: ROTATOR CUFF REPAIR
- TENOTOMY (Experimental): TENOTOMY OF LHBT + ROTATOR CUFF REPAIR
  Interventions: Procedure: ROTATOR CUFF REPAIR

INTERVENTIONS:
Procedure: ROTATOR CUFF REPAIR — ROTATOR CUFF REPAIR

SUMMARY:
The function of the long head of the biceps tendon (LHBT) in the glenohumeral joint generates controversy among researchers. For some, the tendon does not have a significant function in the shoulder, while others consider it acts as a depressor of the humeral head and a stabilizer of the joint. These functions may be enhanced in cases of rotator cuff injuries, where compensatory hypertrophy and/or instability of the LHBT can occur, which can also be a source of pain. One of the imaging techniques used for diagnosing these injuries is ultrasound.

Initially, G. Walch proposed tenotomy of the LHBT in massive rotator cuff tears to improve pain and, in some cases, shoulder function. Currently, many authors advocate tenotomy of the LHBT as an adjunct to rotator cuff repair to avoid postoperative pain. However, there is no evidence that this procedure improves the clinical outcomes of isolated rotator cuff repair.

Based on the pathophysiology of the LHBT associated with rotator cuff injuries and the current trend to perform tenotomies in conjunction with cuff repair, the objectives of this doctoral thesis project were:

To compare the clinical and imaging outcomes of arthroscopic rotator cuff repairs with and without LHBT tenotomy.

To analyze the position and cross-sectional area of the LHBT in the bicipital groove using ultrasound in cases with and without tenotomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years
* Partial supraspinatus tears (≥ 50% thickness)
* Complete supraspinatus tears ≤ 3 cm in the coronal plane
* Muscle atrophy less than stage 2 according to Thomazeau
* Presence of the LHBT in the bicipital groove

Exclusion Criteria:

* Patients younger than 40 or older than 65 years
* LHBT rupture
* Partial supraspinatus tears < 50% thickness
* Supraspinatus tears > 3 cm
* Tears of other rotator cuff tendons, with or without supraspinatus involvement
* Traumatic tears with surgery performed less than 3 months after injury
* Muscle atrophy ≥ stage 2 Thomazeau
* Associated degenerative glenohumeral pathology (> Samilson 1)
* Previous shoulder surgeries
* Previous shoulder infections
* Associated peripheral neurological injuries
* Degenerative neurological conditions
* Patients who refused to sign informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Constant Murley | 24 month
  100-point standardized tool for assessing shoulder function, comprising four domains Pain (0-15 points) daily life activity (0-20 points) range of motion (0-40 points) strenght (0-25 points)
  0 (the worst) - 100 (the best)

SECONDARY OUTCOMES:
ASES | 24 MONTHS
  The ASES score (American Shoulder and Elbow Surgeons score) is a 100-point questionnaire used to assess shoulder function and pain, with a higher score indicating better outcomes.
  From 0 (worst) to 100 (best).
cross sectional area of the LHBT | 24 months
  Ultrasound Imaging: Integrity of the supraspinatus tendon (SST) repair, presence of the long head of the biceps tendon (LHBT) in the bicipital groove (BG), and cross-sectional area of the LHBT at three levels of the BG (proximal, middle, and distal).
  mesured in mm2

IPD SHARING:
Plan to Share IPD: Undecided